CLINICAL TRIAL: NCT03703557
Title: Feasibility Study on the Possibility of Isolation of Volatile Organic Compounds (VOCs) Related to the Olfactory Signature of Breast Cancer
Brief Title: Isolation of Volatile Organic Compounds (VOCs) Related to the Olfactory Signature of Breast Cancer
Acronym: KDOG2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IC 2018-01
Record Dates: First submitted 2018-07-10; First posted 2018-10-12 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Surgery
Keywords: Breast; Volatile organic compounds
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, open, monocentric study with risks and minimal constraints
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sorbstar® (Experimental): Odour sampling: Rub hands with Sorbstar® before and post-surgery
  Interventions: Diagnostic Test: Sorbstar®
- Dog detection (Experimental): Odour sampling: Sleep over a night with a compress on the affected breast before and after surgery
  Interventions: Diagnostic Test: Odour sampling

INTERVENTIONS:
Diagnostic Test: Sorbstar® — Thermodesorption method coupled with full two-dimensional gas chromatography and mass spectrometry.
  Arms: Sorbstar®
Diagnostic Test: Odour sampling — Analyzed by the dogs of Curie Institute at the training centers
  Arms: Dog detection

SUMMARY:
To ascertain the possibilities to isolate the breast cancer olfactive signature.

DETAILED DESCRIPTION:
Patient recruitment during the first surgery consultation in Curie Institute. Odor sampling (non-invasive) with an odor-sensing polymer (Sorbstar® polymer developed especially for the trace level analysis), on:

* The hands, before and after surgical excision of the tumor (friction of the hands)
* The diseased breast, before and after surgical excision of the tumor (via a compress positioned on the breast for 1 night)
* The tumor, during the surgical procedure (odor collection over a tumor sample).

Each patient will be her own witness, before and after surgical excision, in an attempt to isolate the chemical signature tracks of breast cancer. The samples after surgery will be made after healing and before implementation of a treatment (chemotherapy and / or radiotherapy).

ELIGIBILITY:
Inclusion Criteria:

1. Patient received in surgery consultation for an invasive non metastatic breast cancer treated by breast-conserving surgery with axillary or sentinel node dissection
2. Of-Age female patient (over 18 years old)
3. Life expectancy > to 1 year at the inclusion
4. Performance status: 0 or 1 or 2
5. Patient benefiting from the social security
6. Signature informed consent of the study

Exclusion Criteria:

1. Neoplasia in progress or neoplasia history of cancer other than breast to be treated.
2. Wound presence on breasts
3. Male subjects
4. Specified metastatic breast cancer
5. Concomitant medication taken one month before the surgical act (antibiotics, corticoids, anti-diabetics)
6. Persons under guardianship or deprived of liberty
7. Impossibility to submit to the medical monitoring expected by the study for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Ascertain breast cancer olfactive signature (Isolation of volatile Organic Compounds to breast cancer by a sensitive technique with an odor-sensing polymer (Sorbstar®) | 12 months
  Isolation of volatile Organic Compounds to breast cancer by a sensitive technique with an odor-sensing polymer (Sorbstar®) on hands. Friction of the hands according to the protocol before and after surgical excision of the tumor. Sorbstar® analyses will be performed with a thermodesorption method coupled with full two-dimensional gas chromatography and mass spectrometry.

SECONDARY OUTCOMES:
Ascertain breast cancer olfactive signature from the tumor (Isolation of volatile Organic Compounds to tumor breast samples by a sensitive technique with an odor-sensing polymer (Sorbstar®). | 13 months
  During the surgical procedure an odor-sensing polymer (Sorbstar®) over the tumor is placed. Sorbstar® analyzes will be performed with a thermodesorption method coupled with full two-dimensional gas chromatography and mass spectrometry.
Ascertain breast cancer detection by the dogs of Curie Institut | 13 months
  Patients sleep over a night with a compress positioned on the affected breast before and after surgery. The compress will be analyzed by the dogs of Curie Institut (results cancer/not cancer).

CONTACTS AND LOCATIONS:
Overall Officials: Roman ROUZIER, Phd, Principal Investigator — Institut Curie; Isabelle FROMANTIN, Phd, IDE, Study Director — Institut Curie
Locations (1):
- INSTITUT CURIE - Site de Saint Cloud, Saint-Cloud, France